CLINICAL TRIAL: NCT00006259
Title: A Phase II Trial of Radiosurgery Alone for Brain Metastases in Elderly Patients or Patients With Poor Performance Status
Brief Title: Stereotactic Radiation Therapy in Treating Patients With Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Andrew Metzger, MD, Ireland Cancer Center at University Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU3399
Record Dates: First submitted 2000-09-11; First posted 2004-03-08 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Cancer
Keywords: tumors metastatic to brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: stereotactic radiosurgery — Patients undergo stereotactic head frame placement, followed by stereotactic radiosurgery using Gamma Knife, on day 1.

SUMMARY:
RATIONALE: Stereotactic radiation therapy may be able to deliver x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: Phase II trial to study the effectiveness of stereotactic radiation therapy in treating patients who have brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of stereotactic radiosurgery without whole brain radiotherapy in elderly patients or patients with poor performance status who have brain metastases. II. Determine the neurologic function in these patients after receiving this treatment regimen. III. Determine the quality of life in these patients with this treatment regimen.

OUTLINE: Patients undergo stereotactic head frame placement, followed by stereotactic radiosurgery using Gamma Knife, on day 1. Quality of life is assessed one week prior to and one week after treatment, and then at 2, 4, 6, 8, 10, and 12 months. Patients are followed at one week, at 2, 4, 6, 8, 10, and 12 months, every 4 months for one year, and then every 6 months for 3 years.

PROJECTED ACCRUAL: Approximately 52 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patients with 1-4 sites of brain metastases Confirmed by MRI with gadolinium texaphyrin scan within two weeks of study If solitary metastases, diameter must be 40 mm or less If multiple metastases, one site may be greater than 30 mm, while all others must be less than 30 mm No metastases in the brainstem or within 5 mm of optic nerves or chiasm Prior surgical resection of metastases allowed if radiographically visible residual disease No prior cranial radiotherapy Patients must be over 65 years of age OR Over 18 years of age with Karnofsky performance status 40-60% All primary histologies allowed except the following: Lymphomas Leukemia Multiple myeloma Small cell lung cancer Germ cell tumors Extracranial disease allowed

PATIENT CHARACTERISTICS: Age: See Disease Characteristics Performance status: See Disease Characteristics Life expectancy: Not specified Hematopoietic: Hemoglobin greater than 8 g/dL Absolute neutrophil count greater than 1,000/mm3 Platelet count greater than 50,000/mm3 Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior chemotherapy allowed Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Prior or concurrent radiotherapy to noncranial sites allowed Surgery: See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2000-01; Primary Completion 2001-11 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Study the effectiveness of stereotactic radiation therapy in treating patients who have brain metastases. | Quality of life is assessed one week prior to and one week after treatment, and then at 2, 4, 6, 8, 10, and 12 months. Patients are followed at one week, at 2, 4, 6, 8, 10, and 12 months, every 4 months for one year, and then every 6 months for 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Donald C. Shina, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States